CLINICAL TRIAL: NCT03471039
Title: Pituitary Adenylate Cyclase-activating Polypeptide (PACAP27) Headache Properties in Migraine Without Aura Patients
Brief Title: PACAP27 Headache Properties in Migraine Without Aura Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Danish Headache Center (Other)
Responsible Party: Principal Investigator, Hashmat Ghanizada, Principal Investigator, Danish Headache Center
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Health Services Research
Other Study IDs: H-17016232
Record Dates: First submitted 2018-03-01; First posted 2018-03-20 (Actual); Last update posted 2019-01-24 (Actual); Status verified 2019-01

CONDITIONS: Migraine Without Aura
MeSH Terms: conditions — Migraine without Aura | interventions — Pituitary Adenylate Cyclase-Activating Polypeptide; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active (Active Comparator): PACAP-27
  Interventions: Drug: PACAP27
- Placebo (Placebo Comparator): Saline
  Interventions: Drug: Saline

INTERVENTIONS:
Drug: PACAP27 — Infusion of PACAP27 over 20 minutes.
  Arms: Active
Drug: Saline — Infusion of Saline over 20 minutes.
  Arms: Placebo

SUMMARY:
Pituitary adenylate cyclase-activating polypeptide (PACAP) is a signaling molecule, localized in sensory and parasympathetic perivascular nerves fibres. PACAP exists i to functional iso-forms Pituitary adenylate cyclase-activating polypeptide-38 (PACAP38) and PACAP27.

ELIGIBILITY:
Inclusion Criteria:

* Migraine patients meeting International Headache Society (IHS) criteria for migraine without aura of both sexes, 18-60 year, 50-100 kg.

  * Fertile women should use safe contraception. Fertile women do not include hysterectomized women or women who are postmenopausal for at least 2 years. Safe contraception includes either Intra Uterine Device (IUD), birth control pills, surgical sterilization of the woman or depot progestogen.

Exclusion Criteria:

* Tension Type headache for more than 5 days the month on average in the last year.

  * All other primary headaches .
  * Headache later than 48 hours before trial start.
  * Daily intake of any medicine other than oral contraception.
  * Ingestion of any form of medicinal product later than 4 times the plasma half-life substance (on trial day), except for oral contraception.
  * Pregnant or breastfeeding women.
  * Headache on the test day or later than 48 hours prior to administration of trial medicine / placebo
  * Migraine within 5 days before the trial date.
  * Ancestral information or clinical signs of (on the day of inclusion):
* Hypertension (systolic blood pressure> 150 mmHg and / or diastolic blood pressure> 100 mmHg)
* Hypotension (systolic blood pressure <90 mm Hg and / or diastolic blood pressure <50 mmHg)

  * Cardiovascular disease of all kinds, including cerebrovascular disease.
  * Anamnestic or clinical signs of mental illness or abuse.
  * Patients with glaucoma or prostatic hyperplasia
  * Anamnestic or clinical signs of diseases of any kind such as the investigating physician is considered relevant for participation in the trial.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2017-08-30 (Actual); Primary Completion 2018-08-30 (Actual); Study Completion 2018-09-30 (Actual)

PRIMARY OUTCOMES:
Headache Scores | 0-12 hours
  Comparison between PACAP27 and Placebo

SECONDARY OUTCOMES:
Facial blood flow (flushing) | 0-120 mins
  PACAP27 induces facial flushing compare to placebo measured by laser speckle contrast imaging

CONTACTS AND LOCATIONS:
Locations (1):
- Danish Headache Center, Glostrup Municipality, Denmark